CLINICAL TRIAL: NCT05142579
Title: EFFECT OF TWO DIFFERENT ENDOTRACHEAL TUBE DETECTION ON PRESSURE WOUND FORMATION IN INTENSIVE CARE UNIT: A RANDOMIZED CONTROLLED STUDY
Brief Title: EFFECT OF ENDOTRACHEAL TUBE DETECTION ON PRESSURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University Pendik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Alev Genç, M.Sc NURSE, Marmara University Pendik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Marmara EAH-ALEV GENÇ
Record Dates: First submitted 2021-03-30; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Pressure Injury
Keywords: Endotracheal Tube; Endotracheal Tube Holder; Bandage; Intensive Care Unit; Pressure Wound
MeSH Terms: conditions — Pressure Ulcer | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: The 60 patients who made up the sample were assigned 2 groups using a computer program that produced random numbers. For the purpose of the study, the groups were encoded as groups A and B, and each group was tested with two different endotracheal tube detection methods which was applied to the patients in the groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENDOTRACHEAL TUBE HOLDER (Experimental): Endotracheal tube holder was used for endotracheal tube detection of patients in this group.
  Interventions: Other: ENDOTRAKEAL TUBE HOLDER
- BANDAGE (Active Comparator): The bandage was used for endotracheal tube detection of patients in this group.
  Interventions: Other: BANDAGE

INTERVENTIONS:
Other: ENDOTRAKEAL TUBE HOLDER — During this process, the tube detection of endotracheal tube holder was changed every 24 hours, and the tubes were repositioned every 4 hours. On the first day of the study, the oral mucosa of patients in this group was evaluated by the eliers oral evaluation guide.Then, with the Braden pressure wound risk diagnostic scale, patients ' Pressure Wound risk assessment was performed. Patients in this group were monitored for four days for oral pressure wound as of the day they were intubated. During this process, patients ' tube holder was changed every 24 hours and the tube was repositioned every 4 hours. At the end of the fourth day, wound evaluation of patients who developed pressure wounds was performed using the international pressure wound staging system and pressure ulcer Recovery Assessment Scale. In addition, pressure wounds of patients who developed pressure wounds were treated in accordance with the recommendation of a plastic surgeon.
  Arms: ENDOTRACHEAL TUBE HOLDER
Other: BANDAGE — On the first day of the study, the oral mucosa of patients in this group was evaluated by the eliers oral evaluation guide.Then, with the Braden pressure wound risk diagnostic scale, patients ' Pressure Wound risk assessment was performed. Patients in this group were monitored for four days for oral pressure wound as of the day they were intubated. During this process, patients ' tube holder was changed every 24 hours and the tube was repositioned every 4 hours. At the end of the fourth day, wound evaluation of patients who developed pressure wounds was performed using the international pressure wound staging system and pressure ulcer Recovery Assessment Scale.In addition, pressure wounds of patients who developed pressure wounds were treated in accordance with the recommendation of a plastic surgeon.
  Arms: BANDAGE

SUMMARY:
This study was conducted to examine the effect of two different tube detection on pressure wound formation in the intensive care unit. The search was carried out with a total of 60 patients that 30 of 60 them are interventions and 30 of 60 as experiments, who were hospitalized in the anesthesia and reanimation intensive care unit of an Educational Research Hospital. The 60 patients who made up the sample were assigned 2 groups using a computer program that produced random numbers. For the purpose of the study, the groups were encoded as groups A and B, and each group was tested with two different endotracheal tube detection methods which was applied to the patients in the groups. Data from the study were collected using the introductory and clinical features form, the braden pressure wound risk diagnostic scale, the pressure ulcer recovery assessment scale, the international pressure wound staging system, and the eilers oral assessment guide. Patients in both groups were monitored for four days for oral presure injury. During this process, the tube detection of both groups was changed every 24 hours, and the tubes were repositioned every 4 hours. At the end of the fourth day, wound assesments of patients who developed pressure wounds were performed by using the international pressure staging system and the pressure ulcer recovery assessment scale. Relatives of the patients who were scheduled to conduct the study were informed about the study by oral and written and their consent was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18-65
* Must be intubated oratraceal

Exclusion Criteria:

* Oral pressure wounds
* Burns on the face
* Diabetes
* Facial and neck trauma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
BANDAGE | At the end of the 4th day, the wound evaluation of the patients who developed pressure ulcers was made with the International Staging System for Pressure Injuries and The Pressure Ulcer Scale for Healing.
  It was determined that the bandage method was better than the ETT method in terms of both the pressure ulcer risk score difference and the tendency to fall, dislocate or remain stable
ENDOTRACHEAL TUBE HOLDER | At the end of the 4th day, the wound evaluation of the patients who developed pressure ulcers was made with the International Staging System for Pressure Injuries and The Pressure Ulcer Scale for Healing.
  It was determined that the bandage method was better than the ETT method in terms of both the pressure ulcer risk score difference and the tendency to fall, dislocate or remain stable

CONTACTS AND LOCATIONS:
Overall Officials: TÜLİN YILDIZ, PhD, Principal Investigator — Namik Kemal University
Locations (1):
- Marmara University Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No